CLINICAL TRIAL: NCT04736368
Title: Empirical Dietary Inflammatory Pattern (EDIP) Based Dietary Suggestion on Disease Activity and Cerebrovascular Function in Crohn's Disease
Brief Title: Effect of EDIP Based Diet on CD Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDIPstudy
Record Dates: First submitted 2021-01-31; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; EDIP diet; Therapy; Cerebrovascular Function
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: The study design was a single-blinded randomized, parallel assignment clinical trial of CD participants was conducted. Participants were randomized in a 1:1 fashion to either 14-weeks of an EDIP based diet or a normal diet .
Who Masked: Participant
Masking Description: The study design was a single-blinded randomized, parallel assignment clinical trial of The study design was single blind and the participants did not know what diet intervention is being given to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDIP Group (Experimental): CD participants will receive EDIP diet information
  Interventions: Other: EDIP Diet Suggestions
- Control Group (Placebo Comparator): CD participants will be given diet suggestions according to routine experience.
  Interventions: Other: diet guidance

INTERVENTIONS:
Other: EDIP Diet Suggestions — CD participants will receive EDIP diet suggestions after random allocation.
  Arms: EDIP Group
Other: diet guidance — Control group will be given diet guidance according to routine experience under the participant's request.
  Arms: Control Group

SUMMARY:
Crohn's disease is a chronic recurrent systemic inflammatory disease. Studies have shown that meat, dairy products, fiber and vitamin D may affect the risk of Crohn's disease. The relationship between other dietary components and disease activity or recurrence in Chron's disease has not been fully studied. Although the patient's diet will affect the degree of disease activity, there is still no recognized daily diet model for CD patients. At present, the change of intestinal microbiome is considered to be one of the causes of IBD, and this change provides a theoretical basis for diet to reduce the inflammatory response in CD patients through the regulation of microbiome. Food driven inflammation may affect the activity of the disease. Brain-gut axis interaction may play an important role in CD and may have an effect on the cerebrovascular system. The investigators aim to evaluate the effects of Empirical Dietary Inflammatory Pattern (EDIP) based dietary suggestions on disease activity and cerebrovascular function as well as changes of intestinal flora and its metabolites amongst Chron's disease participants of all ages.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic recurrent systemic inflammatory disease, mainly affecting the gastrointestinal tract, accompanied by extra-intestinal complications and immune dysfunction. The relationship between other dietary components and disease activity or recurrence has not been fully studied and there is still no recognized daily diet model for CD. At present, the change of intestinal microbiome is considered to be one of the causes of Irritable Bowel Disease (IBD), and this change provides a theoretical basis for diet to reduce the inflammatory response those with CD through the regulation of microbiome. In inflammatory diseases, the potential inflammation of food may affect the activity of the disease. Empirical Dietary Inflammatory Pattern (EDIP) is a dietary inflammation index based on food group. 18 food groups were selected to evaluate the levels of inflammatory factors in human body which have already been verified by two independent female and male cohorts. The construction and validation of the scoring model revealed a strong correlation between EDIP and three plasma inflammatory markers: IL-6, CRP and TNFaR2, as well as other markers, such as adiponectin and the overall inflammatory marker score. Therefore, EDIP can be derived in a standardized way in different populations and be used to examine association with diseases whose pathogenesis is mainly attributed to chronic inflammation. Dietary inflammation index (DII) is a previously developed inflammation index based on nutrients. Compared to DII, dietary patterns based on food groups, such as EDIP, are more valuable for the establishment of dietary guidelines for health promotion and disease prevention. In addition, the brain-gut axis is the kink between the central nervous system and intestinal function but has not been extensively studied. In view of the fact that autoimmune diseases, and brain-gut axis interaction may play an important role in CD, we speculate that cerebrovascular function may also change during the occurrence and development of CD, especially during the EDIP score-based diet. The investigators plan to carry out a randomized controlled trial to systematically study the effects of EDIP score-based dietary suggestions on disease activity and cerebrovascular function of CD patients, as well as the changes of intestinal flora and its metabolites. The primary aim of this study is to systematically study the effects of EDIP based dietary recommendations on disease activity and cerebrovascular function of CD patients and establish a diet model suitable for CD patients. The secondary aims are to explore the possible changes of intestinal flora and its metabolites, and evaluate the changes of cerebrovascular function and the possible mechanism of their actions on CD.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed diagnosis of CD were actively included for different treatment strategies.

Exclusion Criteria:

* Participants with multi-system organ failure and/or other severe diseases not suitable for CD treatment intervention were further excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-26 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Chron's Disease Activity Index | 14 weeks post enrollment.
  The participants disease activity will be assessed with CDAI index.

SECONDARY OUTCOMES:
Mucosal Changes | 14 weeks post enrollment.
  The status and degree of mucosal healing will be assessed by colonoscopy.
Cerebrovascular Function | 14 weeks post enrollment.
  Near infrared spectroscopy will be used to assess cerebrovascular function.